CLINICAL TRIAL: NCT01716403
Title: Influence of Telaprevir Exposure on the Severe Anemia Induced by Ribavirin/Pegylated Interferon/Telaprevir Tri-therapy in HCV Infected Patients
Brief Title: Telaprevir Exposure and Severe Anemia in HCV Infected Patients Treated by Tri-therapy
Acronym: Ribatela
Status: Terminated | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 1211
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: C Hepatitis, Tri Therapy
Keywords: C hepatitis, telaprevir concentration, ribavirin oncentration, anemia
MeSH Terms: conditions — Hepatitis C; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV tritherapy and anemia: HCV-genotype 1 infected patients
  Interventions: Biological: Diagnostic: protocol designed to evaluate one or more interventions aimed at identifying a disease or health condition

INTERVENTIONS:
Biological: Diagnostic: protocol designed to evaluate one or more interventions aimed at identifying a disease or health condition

SUMMARY:
The risk of severe anemia is increased in patients treated by tri-therapy compared to patients treated by bitherapy. The underlying mechanisms involved in this toxicity remain unexplored but could also depend on the global exposure of telaprevir. The trough concentration or AUC of telaprevir could therefore be a predictive factor of the onset of anemia in patients treated by ribavirin/PEG-INF/telaprevir. The early measurement of telaprevir and ribavirin concentrations could help to manage HCV tri-therapy to improve tolerance and SVR.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman older than 18 yr. 2- HCV genotype 1 infection as confirmed by a positive viral load 6 months after the selection visit or confirmed by the mean of a liver biopsy within 1 year before screening for the study.

  3- Patient with one of the following criteria: Patient naive of any treatment against HCV infection Or Prior null responder patient: patient previously treated by ribavirin/PEG-INF for at least 12 weeks and whom HCV viral load decline was <2 log at week 12 Or Prior partial responder patient: patient previously treated by ribavirin/PEG-INF for at least 12 weeks, who never had a negative viral load while the viral load decline was >2 log at week 12 Or Prior relapser patient: patient previously treated by ribavirin/PEG-INF for 48 weeks, with a negative viral load at the end of treatment and a positive viral load 6 months later 4- Patient who has stopped his treatment for at least 12 weeks 5- Patient who had a liver biopsy or a Fibroscan within the 24 months before the start of the study with a Metavir fibrosis score F ≥ 3.

  6- Patient who fulfills criteria for telaprevir treatment as defined by the licence 7- Patients who accepts to use 2 contraceptive methods until 6 months after the end of the treatment 8- Patient who had given his written informed consent 10- Patient insured under the french social security system

Exclusion Criteria:

1- Infection/co-infection by HCV genotype different than genotype 1 2- Patient with a medical contraindication to PEG-INF or ribavirin 3- Patient with history of allergy or intolerance to telaprevir 4- Patient using contraindicated drugs 5- Patient with history of decompensated liver disease and/or presenting biochemical measurements as follows at the inclusion visit:

* International Normalized Ratio (INR) > 1,5
* Albumin <3,3 g/dl
* Total bilirubin>1,8 N apart for patient with Gilbert syndrome 6- Liver disease from other causes 7- Patient with hepatocellular carcinoma or history of cancer 8- Patient with a history of graft transplantation and treated by immunosuppressive drugs 9- Patient who are regularly treated by corticosteroids 11- Patient with hemophilia or coagulation troubles 12- HIV or HBV co-infection 14- Patient with body mass index> 30 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 48 HCV-genotype 1 infected patients (16 naive patients, 16 prior partial responders/relapsers and 16 prior null responders to ribavirin/PEG-INF treatment)
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
telaprevir concentration and area under the curve | Day 0, Day 2, week 2, week 4, week 8 and week12

SECONDARY OUTCOMES:
ribavirin concentration and area under the curve | Day 0, Day 2, week 2, week 4, week 8 and week12

OTHER OUTCOMES:
viral load | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Zarski, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France